CLINICAL TRIAL: NCT01372839
Title: The Safety and Efficacy of Intensive Statin Therapy in PCI Patient With Acute Coronary Syndrome
Brief Title: Intensive Statin Therapy in PCI Patient With Acute Coronary Syndrome
Acronym: PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Ling Tao, Department of Cardiology of Xijing Hospital; Fourth Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xj050511
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2010-07

CONDITIONS: Myocardial Infarction; Unstable Angina
Keywords: Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator): 80mg/d ×2d before PCI. After PCI, atorvastatin 40mg/d until 30 days later, and then followed by usual care
  Interventions: Drug: Atorvastatin
- Usual care (Other): statin dose should not be higher than that described in exclusion criteria.
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80mg/d ×2d before PCI. After PCI, atorvastatin 40mg/d until 30 days later, and then followed by usual care
  Arms: Atorvastatin
Drug: Statin — Usual care, but statin dose should not be higher than that described in exclusion criteria
  Arms: Usual care

SUMMARY:
Compare with regular regimen, the aim of this study is to testify whether having more statin during PCI will benefit in Chinese population, and to find out optimal dose of the drug for patient after PCI.

DETAILED DESCRIPTION:
This study is designed to find out whether patients undergoing PCI can benefit from intensive atorvastatin treatment compared with routine treatment on chinese population.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old
* Patients with clinical diagnosis of ACS
* Evidence of a personally signed and dated informed consent document

Exclusion Criteria:

* Taking or, needing to take atorvastatin over than 20mg/d or any other equivalent statin in the next 6 months, or needing to take fibrates simultaneously according to investigators' judgment.
* LDL-C < 1.8mmol/L in patients without statin therapy in 1 months
* Endstage congestive heart failure, or LVEF < 30%
* Active hepatic disease or hepatic dysfunction, or AST/ALT > 1.5UNL
* Myopathy or increased creatine kinase (CK>2 UNL)
* Severe renal dysfunction(Scr > 3 mg/dl or 264μmol/L)
* Allergic or experienced serious adverse reaction to HMG-CoA reductase, or ineligible to take statin as investigator's judgment
* Severe aortic valve stenosis or severe mitral stenosis, Obstructive hypertrophic cardiomyopathy, pericardial diseases
* Pregnancy, lactation, or child bearing potential women without any effective contraception
* Accompanied with malignant disease or other disease, which cause life expectancy < 6 months
* Participating in other interventional clinical trails using drugs or devices
* Patients with any condition which, in the investigator's judgment, might increase the risk to the subject for any adverse event or abnormal laboratory finding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
30-day major adverse cardiovascular events (combined endpoints of cardiac death, myocardial infarction, and target vessel revascularization ) after PCI | 30-day

SECONDARY OUTCOMES:
Post-procedural change of inflammatory biomarkers (hs-CRP) | 24h
Morbidity of CIN | 48h
Elevation of ALT, AST and CK | 6 months
  Proportion of patients who experience at least once AST>3UNL，ALT>3UNL or CK>5UNL after initiation of study treatment. Proportion of patients who experience at least once AST, ALT, or CK>UNL after initiation of study treatment.
Number of Participants with Adverse Events | 6 months
  Proportion of patients who take reduced dose of atorvastatin, withdraw study treatment, or withdraw study due to adverse events
Combined endpoint of MACEs, cardiac hospitalization and cerebrovascular events | 6 months
  Combined endpoint of death, cardiac death, myocardial infarction, heart failure, cardiac hospitalization, revascularization, and cerebrovascular events within 6 months after PCI.
serum adiponectin concentration | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Study Director — Division of Cardiology, Peking University First Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China